CLINICAL TRIAL: NCT06375304
Title: Antiretroviral Speed Access Program Switch Study (The ASAP Switch Study) - A Pilot Study to Switch ART-experienced and Newly-referred Migrant People With HIV to B/F/TAF
Brief Title: The Antiretroviral Speed Access Program Switch (ASAP-Switch) Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Bertrand Lebouche, Clinician Scientist and associate professor of medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-37-2024-10384
Record Dates: First submitted 2024-04-12; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
Keywords: HIV; multidisciplinary model of care; patient-reported experiences; patient-reported outcomes; switch
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Antiretroviral Speed Access Program Switch (Other): HIV (type 1) infected adults born outside of Canada (migrants) and recently moved to province of Quebec (less than 2 years), ART-experienced, newly referred at the study sites.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — The intervention consists of prescribing B/F/TAF to eligible ART-experienced migrant patients, free of charge, in four care settings, for 12 months (48 weeks).
  B/F/TAF is a fixed-dose combination of bictegravir (50 mg), emtricitabine (200 mg), and tenofovir alafenamide (25 mg), administered orally, once daily, without food requirements.

SUMMARY:
This project builds on our experience with the ASAP Study (McGill University Health Centre research ethics board: MP-37-2020-4911). The goal of this study is to better understand the experience of migrant people with Human Immunodeficiency Virus (HIV) of having their treatment switched to Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF). In other words, the investigators want to evaluate how feasible and acceptable this switch is, and how participants will take B/F/TAF (fidelity) and remain on it. The investigators also want to know more about migrant people with HIV's experience of care; namely, how often they see their HIV specialist or other healthcare professionals, and their healthcare coverage (the type of insurance that they have).

DETAILED DESCRIPTION:
International migrants represent an increasing portion of people with HIV in Canada. Making sure migrant people with HIV have access to treatment and care is crucial for their health and wellbeing. It is also important to make sure that they have a good experience of care and treatment. Several treatments exist for HIV, and many migrant people with HIV arrive in Quebec with a current or past experience of taking an HIV treatment. Sometimes, it is a treatment that cannot be continued here, for different reasons. Thus, their treatment must be 'switched', that is, changed to another treatment more affordable, simpler, or more efficient.

B/F/TAF is one HIV treatment. B/F/TAF is simple to take (one small-sized pill a day), safe, highly effective for almost all people with HIV, and ideal when one switches from one treatment to another. If participants take part in this study, their treatment will be switched to B/F/TAF; it will be provided free of charge for the participants.

The goal of this study is to better understand the experience of migrant people with HIV of having their treatment switched to B/F/TAF. In other words, the investigators want to evaluate how feasible and acceptable this switch is, and how participants will take B/F/TAF (fidelity) and remain on it. The investigators also want to know more about migrant people with HIV's experience of care; namely, how often they see their HIV specialist or other healthcare professionals, and their healthcare coverage (the type of insurance that they have).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand the requirements of study participation and provide signed and dated written informed consent prior to performing study procedures;
* 18 years of age or older;
* Living with HIV (type 1) (as confirmed by a fourth generation HIV Ag/Ab combination assay);
* Patients at their first visits ever at the study site;
* Born outside of Canada, and arrived in the province of Quebec from another province or country to reside temporarily or permanently in the last 24 months;
* ART-experienced, that is, with past or current experience of taking ART to treat HIV, with or without treatment interruption(s) for any clinical or personal reason;
* Individuals assigned female at birth may be eligible to enter and participate in the study in the following circumstances:

  * is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy, or bilateral oophorectomy or,
  * is of child-bearing potential with a negative pregnancy test at Screening (& baseline visit) and reporting no plans to become pregnant in the next year.

Patients with documented historical resistance to HIV-1 reverse transcriptase inhibitors will be eligible, including: M184I/V alone or in combination with up to 2 thymidine analogue-associated mutations (TAMs) (M41L, D67N, K70R, L210W, T215F/Y, or K219Q/E/N/R).

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant;
* Current alcohol or substance use judged by the investigator to potentially interfere with participant study compliance;
* Active tuberculosis infection;
* Acute hepatitis < 30 days before enrollment;
* Known hypersensitivity to B/F/TAF, its metabolite or formulation excipient;
* Documented or suspected resistance to integrase inhibitors as per clinical judgment (e.g., history of poor adherence and/or poor virological control on an InSTI-based regimen);
* Documented multi-NRTI resistance mutations/substitutions: K65R/N/E, T69 insertion, or 3 or more TAMs (M41L, D67N, K70R, L210W, T215F/Y, K219E/Q);
* Any of the following laboratory values at screening:

  * Alkaline Phosphatase>3 × ULN
  * aspartate aminotransferase (AST) >5 × upper limit of normal
  * alanine aminotransferase (ALT) >5 × upper limit of normal
  * Hemoglobin<8.0 g/dL
  * Estimated creatinine clearance (CrCL) ≤30 mL/min/1.73 m2 based on the Cockcroft-Gault equation for creatinine clearance (CLcr)
  * Platelets< 50,000/mm3
* Participation or planned participation in any other clinical study (including observational studies) without prior approval from the sponsor;
* Any reason, in the opinion of the investigator, which would make the candidate inappropriate for participation in an investigative study involving oral medications (e.g., inability to understand the study information leaflet, to provide written consent);
* Concomitant use of drugs with contraindication or drug-drug interactions with B/F/TAF;
* Active malignancy requiring acute systemic therapy;
* History of or current clinical decompensated liver cirrhosis (e.g., ascites, encephalopathy, or variceal bleedings).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the switch | within 7 days of first clinic visit
  Feasibility refers to the extent to which an implementation target can be successfully used or deployed within a given setting. The investigators will measure what percentage of participants have done the switch and what percentage have not done the switch. For the rapid switch, the investigators will use a threshold of 75% achieving rapid switch (i.e., within 7 days of first clinic visit). Therefore, the investigators will report the percentage that achieved the switch within 7 days.
Acceptability | From baseline to week 48.
  Acceptability refers to the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. The investigators will assess the acceptability of: rapidity, the treatment being free-of-charge for patients, and the regimen choice. It will be measured with the 4-item Acceptability of Intervention Measure (AIM), using the following thresholds:
  * ≥M*=4/5 for acceptability of rapid treatment;
  * ≥M=4/5 for acceptability of free treatment.
acceptability of the regimen | From baseline to week 48.
  After initiation, acceptability of the regimen choice will be assessed using the ACCEptance by the Patients of their Treatment (ACCEPT©) questionnaire, including the 3-item 'General acceptance' subscale and the 5-item 'Acceptability of side effects' subscale:
  • ≥M=4/5 for acceptability of the new ART regimen (in general and concerning its side effects).
  The response options range from 1 = "completely disagree" (worst or least acceptable) to 5 = "completely agree" (best or most acceptable).
Acceptability of the intervention | From baseline to week 48.
  Acceptability of the intervention as a whole will also be assessed in terms of readiness with a 2-item readiness measure and a measure of treatment self-efficacy with thresholds of:
  * ≥M=8/10 indicating readiness to start the new regimen (i.e., B/F/TAF);
  * ≥M=16/20 indicating treatment self-efficacy.
    * M: Mean or average.
  The responses are on a scale from 0 to 10 (10 being the best or most acceptable).
Fidelity | From enrolment to week 72.
  Fidelity concerns the degree to which a program is delivered as intended. It will be evaluated with thresholds of:
  • ≥80% for study visit attendance;
  ≥90% for self-reported regimen adherence in the past 30 days and in the last 7 days.

SECONDARY OUTCOMES:
ART initiation (HIV care cascade milestones) | From enrolment to baseline.
  o Treatment (ART) initiation: Proportion and/or time in days to attaining (or maintaining, as relevant).
Viral suppression (HIV care cascade milestones) | From enrolment to week 72 or until viral suppression happens (whichever comes first).
  o Viral suppression (HIV viral load < 50 copies/mL): Proportion and/or time in days to attaining (or maintaining, as relevant)
Retention in HIV care (HIV care cascade milestones) | From enrolment to week 48.
  o Retention in HIV care (i.e., at least 1 clinic visit with a physician per 6-month period of study participation; i.e., a minimum of two visits in total including one within the first 6 months and one within the last 6 months of the first 12 months of the study, with a buffer time period of +/- 6 weeks).
consultations at the study site (Nature of clinical pathways) | From enrolment to week 72.
  o Occurrence and frequency of consultations with healthcare professionals from different disciplines (e.g., physician, pharmacist, nurse, social worker, psychologist, psychiatrist) at the study site.
consultations at other care centres or organizations (Nature of clinical pathways) | From enrolment to week 72.
  o Self-reported occurrence and frequency of consultations at other care centres or organizations.
healthcare coverage | From enrolment to week 72.
  Identification and changes of the type of medical coverage for HIV received by participants as mentioned on patient health records. For example, a change in healthcare coverage from the Interim Federal Health Program to the Régie de l'assurance maladie du Québec (RAMQ), along with the percentages of coverage for the participants' treatment will be noted and recorded by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lebouché, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada